CLINICAL TRIAL: NCT00509392
Title: Radiofrequency Endovenous ClosureFAST vs. Laser Ablation for the Treatment of Great Saphenous Reflux: A Multicenter, Single-Blinded, Randomized Study (RECOVERY)
Brief Title: ClosureFAST vs. Laser Ablation for the Treatment of GSV Disease: A Multicenter, Single-Blinded, Randomized Study.
Acronym: RECOVERY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Collaborators: VNUS Medical Technologies, A Covidien Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CVL-06-03
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Venous Reflux
Keywords: Varicose veins, venous reflux, GSV disease
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seg. RF Ablation & ClosureFAST catheter (Active Comparator): Seg. RF Ablation & ClosureFAST catheter
  Interventions: Device: Seg. RF Ablation & ClosureFAST catheter
- Endovenous Laser (Active Comparator): Treatment invention of venous disease with an Endovenous Laser.
  Interventions: Device: Endovenous Laser

INTERVENTIONS:
Device: Seg. RF Ablation & ClosureFAST catheter — Seg. RF Ablation & ClosureFAST catheter
  Other Names: VNUS
  Arms: Seg. RF Ablation & ClosureFAST catheter
Device: Endovenous Laser — laser catheter
  Other Names: Commercially approved laser catheter systems.
  Arms: Endovenous Laser

SUMMARY:
The objective of this post-market study is to compare the post-procedure recovery between two types of minimally invasive catheter treatments for venous disease in the Great Saphenous Vein.

DETAILED DESCRIPTION:
Comparison of the post-procedure recovery of radiofrequency (RFA) treatment vs. laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must provide written informed consent.
* Must be a candidate for either treatment with Radiofrequency Ablation (RFA) or endovenous laser.

Exclusion Criteria:

* Subjects who require additional treatments in either leg within 30 days before or after the study procedure.
* Subjects who are participating in another investigational study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lian Cunningham, MD, Study Director — VNUS Medical Technologies, A Covidien Company
Locations (1):
- Oregon Health Sciences, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Almeida JI, Kaufman J, Gockeritz O, Chopra P, Evans MT, Hoheim DF, Makhoul RG, Richards T, Wenzel C, Raines JK. Radiofrequency endovenous ClosureFAST versus laser ablation for the treatment of great saphenous reflux: a multicenter, single-blinded, randomized study (RECOVERY study). J Vasc Interv Radiol. 2009 Jun;20(6):752-9. doi: 10.1016/j.jvir.2009.03.008. Epub 2009 Apr 22. PMID 19395275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from March - December 2007. Medical offices/clinics and university hospital.
Units Other Than Participants: limbs
Groups:
- Radiofrequency (RF) Ablation: Radiofrequency (RF) thermal ablation using the ClosureFAST (CLF) RF Catheter (VNUS Medical Technologies, San Jose, CA)
- Endovenous Laser (EVL) Ablation: Endovenous Laser (EVL) ablation with a 980-nm laser (Biolitec, East Longmeadow, MA)
- RF / EVLA: Bilateral treatment where one limb is treated with RFA and the contralateral limb is treated with EVL
Period: Overall Study
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation | RF / EVLA
Started | 32; 42 limbs | 33; 37 limbs | 4; 8 limbs
Completed | 32; 42 limbs | 33; 37 limbs | 4; 8 limbs
Not Completed | 0; 0 limbs | 0; 0 limbs | 0; 0 limbs

BASELINE CHARACTERISTICS:
Population: 69 subjects were enrolled and 87 limbs were treated. There were 4 enrolled subjects that had bilateral treatment where one limb was treated with RF and the other limb was treated with EVL. To account for this, 2 subjects were added to the total number of baseline RF participant group and 2 were added to the baseline EVL participant group.
Units Other Than Participants: limbs
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation | Total
Number analyzed (Participants) | 34 | 35 | 69
Number analyzed (limbs) | 46 | 41 | 87
Age, Categorical [Count of Units; unit: limbs]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 30 | 70
  >=65 years | 6 | 11 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (12.8) | 52.4 (15.3) | 52.37 (15.3)
Sex: Female, Male [Count of Units; unit: limbs]
  Female | 38 | 31 | 69
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: limbs]
  United States | 25 | 23 | 48
  Germany | 21 | 18 | 39
VCSS [Mean (Standard Deviation); unit: Scores on a scale] — Venous Clinical Severity Score (0-30 total overall score):
  0(minimum)- No evidence of venous disease 30(maximum)- Severe venous disease
  Scores on a scale | 4.7 (3.1) | 4.9 (2.8) | 4.8 (3.0)
CEAP [Number; unit: limbs] — Clinical/Etiology/Anatomy/Pathophysiology Score
  CEAP Class 2: Clinical classification for individuals with varicose veins
  limbs
    CEAP Class 2 | 43 | 36 | 79
    Not CEAP Class 2 | 3 | 5 | 8
CIVIQ [Mean (Standard Deviation); unit: Score on a questionnaire] — Chronic Venous Insufficiency Questionnaire(CIVIQ) for Quality of Life (QOL). (Min 20- Max 100).
  Global index and an outline of 4 quality-of-life dimensions-"pain" (4 items), "physical" (4 items), "psychological" (9 items), and "social" (3 items). A low global (total) score corresponds to greater patient comfort.
  Score on a questionnaire | 40.6 (17.2) | 40 (14.5) | 40.3 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Pain 0-10 scale (10 most severe)
Time Frame: 48 Hour
Population: Data available at 48 hr follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 46 | 41
units on a scale | 0.7 (0.9) | 1.9 (1.6)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Pain
Description: Pain 0-10 scale (10 most severe)
Time Frame: 1 Week
Population: Data available at 1-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 40 | 36
units on a scale | 0.2 (0.6) | 1.8 (1.8)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Primary Outcome: Pain
Description: Pain 0-10 scale (10 most severe)
Time Frame: 2 Weeks
Population: Data available at 2-week follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 43 | 39
units on a scale | 0.1 (0.4) | 1.2 (1.7)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Primary Outcome: Pain
Description: Pain 0-10 scale (10 most severe)
Time Frame: 1 Month
Population: Data available at 1 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 46 | 41
units on a scale | 0.2 (0.8) | 0.4 (1.2)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.2962, t-test, 2 sided

5. Primary Outcome: Tenderness
Description: Tenderness 0-10 scale (10 most severe)
Time Frame: 48 Hour
Population: Data available at 48hr visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 46 | 41
units on a scale | 0.9 (1.3) | 2.0 (2.3)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0048, t-test, 2 sided

6. Primary Outcome: Tenderness
Description: Tenderness 0-10 scale (10 most severe)
Time Frame: 1 Week
Population: Data available at 1-week follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 40 | 36
units on a scale | 0.5 (1.2) | 1.6 (1.8)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0036, t-test, 2 sided

7. Primary Outcome: Tenderness
Description: Tenderness 0-10 scale (10 most severe)
Time Frame: 2 Weeks
Population: Data available at 2-week follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 43 | 39
units on a scale | 0.3 (0.7) | 1.2 (1.5)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0005, t-test, 2 sided

8. Primary Outcome: Tenderness
Description: Tenderness 0-10 scale (10 most severe)
Time Frame: 1 Month
Population: Data available at 1 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 46 | 41
units on a scale | 0.3 (1.0) | 0.5 (1.2)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.5761, t-test, 2 sided

9. Primary Outcome: Ecchymosis
Description: 0-5 scale (5 most severe) 0: None
  1. <25%
  2. 25-50%
  3. 50-75%
  4. 75-100%
  5. Above or below treated (tx) segment
Time Frame: 48 Hours post treatment (no baseline)
Population: Data available at 48hrs follow-up visit
Measure: Number; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 45 | 41
limbs
  0 | 30 | 8
  1 | 15 | 13
  2 | 0 | 14
  3 | 0 | 5
  4 | 0 | 1
  5 | 0 | 0
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p < 0.0001, Fisher Exact

10. Primary Outcome: Ecchymosis
Description: 0-5 scale (5 most severe) 0: None
  1. <25%
  2. 25-50%
  3. 50-75%
  4. 75-100%
  5. Above or below tx segment
Time Frame: 1 Week post treatment (no baseline)
Population: Data available at 1-week follow-up visit
Measure: Number; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 40 | 35
limbs
  0 | 26 | 9
  1 | 13 | 12
  2 | 0 | 10
  3 | 1 | 4
  4 | 0 | 0
  5 | 0 | 0
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p < 0.0001, Fisher Exact

11. Primary Outcome: Ecchymosis
Description: 0-5 scale (5 most severe) 0: None
  1. <25%
  2. 25-50%
  3. 50-75%
  4. 75-100%
  5. Above or below tx segment
Time Frame: 2 Weeks post treatment (no baseline)
Population: Intent to treat/ SP: Data available at 2-week follow-up visit
Measure: Number; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 43 | 39
limbs
  0 | 35 | 13
  1 | 7 | 18
  2 | 1 | 6
  3 | 0 | 2
  4 | 0 | 0
  5 | 0 | 0
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p < 0.0001, Fisher Exact

12. Primary Outcome: Ecchymosis
Description: 0-5 scale (5 most severe) 0: None
  1. <25%
  2. 25-50%
  3. 50-75%
  4. 75-100%
  5. Above or below tx segment
Time Frame: 1 Month post treatment (no baseline)
Population: Data available at 1- month follow-up visit
Measure: Number; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 46 | 40
limbs
  0 | 45 | 31
  1 | 1 | 9
  2 | 0 | 0
  3 | 0 | 0
  4 | 0 | 0
  5 | 0 | 0
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0050, Fisher Exact

13. Primary Outcome: Complications
Description: Sequelae at any follow-up
Time Frame: 1 month
Population: Data up to one month follow up visit
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 46 | 41
limbs
  Hyperpigmentation | 1 | 0
  Phlebitis | 0 | 8
  Paresthesia | 2 | 3
  Erythema | 0 | 6
  Infection | 0 | 0
  Thrombus Extention (TE)/Deep Vein Thrombosis (DVT) | 0 | 3

14. Secondary Outcome: VCSS
Description: Venous Clinical Severity Score (0-30 total overall score):
  0(minimum)- No evidence of venous disease 30(maximum)- Severe venous disease
Time Frame: 48 Hours
Population: Data at 48 hours for follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 46 | 41
units on a scale | 4.7 (1.6) | 6.2 (2.5)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0009, t-test, 2 sided

15. Secondary Outcome: VCSS
Description: as for outcome 14
Time Frame: 1 Week
Population: Data at 1-week follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 40 | 35
units on a scale | 4.2 (1.5) | 5.9 (2.3)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

16. Secondary Outcome: VCSS
Description: as for outcome 14
Time Frame: 2 Weeks
Population: Data at 2 week follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 43 | 39
units on a scale | 4.0 (1.8) | 5.3 (1.9)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0035, t-test, 2 sided

17. Secondary Outcome: VCSS
Description: as for outcome 14
Time Frame: 1 Month
Population: Data at 1- month follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 46 | 41
units on a scale | 2.7 (2.2) | 3.2 (1.8)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.2825, t-test, 2 sided

18. Secondary Outcome: Change in CIVIQ QOL
Description: Chronic Venous Insufficiency Questionnaire(CIVIQ) for Quality of Life(QOL). (Min 20- Max 100).
  Global index and an outline of 4 quality-of-life dimensions: "pain" (4 items), "physical" (4 items), "psychological" (9 items), and "social" (3 items). A low global (total) score corresponds to greater patient comfort.
  Change from Baseline
Time Frame: 48 Hours
Population: Data at 48 hrs follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 44 | 40
units on a scale | -13.5 (14.6) | -7.1 (19.0)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0854, t-test, 2 sided

19. Secondary Outcome: Change in CIVIQ QOL
Description: as for outcome 18
Time Frame: 1 Week
Population: Data at one week follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 33 | 35
units on a scale | -19.1 (13.9) | -9.4 (13.3)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0044, t-test, 2 sided

20. Secondary Outcome: Change in CIVIQ QOL
Description: Chronic Venous Insufficiency Questionnaire(CIVIQ) for Quality of Life(QOL) (Min 20- Max 100).
  Global index and an outline of 4 quality-of-life dimensions: "pain" (4 items), "physical" (4 items), "psychological" (9 items), and "social" (3 items). A low global (total) score corresponds to greater patient comfort.
  Change from Baseline
Time Frame: 2 Week
Population: Data at 2-week follow up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 40 | 36
units on a scale | -19.9 (14.7) | -12.4 (17.6)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.0457, t-test, 2 sided

21. Secondary Outcome: Change in CIVIQ QOL
Description: as for outcome 18
Time Frame: 1 Month
Population: Data at 1 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: limbs
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Number analyzed (Participants) | 34 | 35
Number analyzed (limbs) | 43 | 39
units on a scale | -17.8 (15.4) | -17.5 (15.2)
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation vs Endovenous Laser (EVL) Ablation; Test type: Superiority or Other; p = 0.9463, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 Month
Description: Number of subjects at risk = Number of subjects with adverse event information
Arm/Group | Radiofrequency (RF) Ablation | Endovenous Laser (EVL) Ablation
Serious Adverse Events (participants affected / at risk) | 0/46 | 1/41
Other Adverse Events (participants affected / at risk) | 2/46 | 9/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency (RF) Ablation (N=46) | Endovenous Laser (EVL) Ablation (N=41)
Thrombus extension (TE) into Common Femoral Vein (CFV) (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency (RF) Ablation (N=46) | Endovenous Laser (EVL) Ablation (N=41)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 6
Paresthesia (Nervous system disorders) | 1 (1) | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data/info related to Study are legal property of VNUS & can be used by PI for publication, communication or scientific presentation only after duly informing VNUS of proposed dissemination, providing to VNUS for review/comment a copy of said proposed publication, communication or scientific presentation & allowing at least 30 days from the time of receipt by VNUS for VNUS to provide comment on said proposed publication, communication or scientific presentation prior to said dissemination.